CLINICAL TRIAL: NCT06909435
Title: Nylon Clip Wear and Patient Perception in Implant Retained Mandibular Overdenture Using PEEK Versus Metal Bar :One Year Randomized Clinical Study
Brief Title: Nylon Clip Wear Assessment in Implant
Acronym: bar implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Amr Heshmat, Associate professor ,Cairo university ,Faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: esthetic committee 49-7-32
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-01

CONDITIONS: Dental Implant Overdenture; Complete Edentulous Patient
Keywords: implant; bar attachment; nylon clip; wear; overdenture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEEK bar (Sham Comparator): Peek bar attachment with Nylon clip for retaining overdenture
  Interventions: Other: PEEK dental bar
- Metal bar (Sham Comparator): metal bar attachment to retain implant overdenture
  Interventions: Other: Metal bar attachment

INTERVENTIONS:
Other: PEEK dental bar — the master stone cast is scanned with external desktop scanner to produce an STL (Standard Tesellation Language) file for a virtual model using the CAD/CAM software (Medit 500i.). The design of the multiunit abutment and bar (Rhein Bar )was selected from the library of the CAD software. The bar dimensions were selected according to the study bar design .
  After the data acquisition, the STL file was imported to the CAM part of the CAD/CAM system to mill PEEK bar from biological high-performance polymer (Bio-HPP) (BreCAM. BioHPP, Bredent GmbH & Co.KG, Senden, Germany) block PEEK type. Multi-unit abutments were screwed to the implants and the PEEK bar was screwed to the abutments .
  Arms: PEEK bar
Other: Metal bar attachment — Co-Cr metal bar group, in the master cast , the multiunit abutment were attached to the implant analogues and plastic abutments were adjusted , prepared and then wax pattern coping was customized on each abutment and was connected to a preformed castable bar 2.4mm Height, (Rhein 83) The bar was placed to be away from the anterior ridge by about 2-3 mm for proper hygiene measures. The wax pattern was then sprued and casted into cobalt- chromium alloy.
  Arms: Metal bar

SUMMARY:
This study is aimed to compare the wear of nylon caps and patient satisfaction in two-implant overdentures with metal bar and Peek bar overlays in the premolar area:

This prospective clinical trial will involve 14 edentulous patients who will receive two implants in the premolar area. Patients will be randomly assigned to two groups: Group A will receive metal bar overlays, and Group B will receive Peek bar overlays. The patients will be evaluated at baseline,one month ,6 month and 12 month The following parameters will be evaluated:

1. Wear of nylon cap: The wear of the nylon cap will be evaluated using a digital microscope at each follow-up visit.
2. Patient satisfaction: Patients will be asked to rate their satisfaction with the overdentureResults: Metal group showed significantly higher roughness and volumetric changes than PEEK regarding baseline, after 3 months, after 6 months, and after 9 months. and there was insignificant difference between them after 12 months as P=0.11.Patient satisfaction scores were significantly higher in the PEEK group, particularly in retention, stability, comfort, and speech domains at both six months and one year (p = 0.04). on a visual analogue scale (VAS) at each follow-up visit.

DETAILED DESCRIPTION:
Forty-six individuals were diagnosed at the outpatient clinic of Removable prosthodontic department at Cairo university and MTI university. From this group, 20 completely edentulous participants of both males and females aged 50 to 60 years were selected based on specific inclusion and exclusion criteria. Each participant provided written consent before this study used their treatment-related radiography data. Ethics committee approval for the study was obtained from the Research Ethics Committee (REC) of the Faculty of Dental Medicine Cairo University, with the reference number REC (No 94/23). The implemented radiation protection methods were in accordance with established guidelines.

Patient selection All the patient involved in the study, they should have inclusion criteria as good bone quantity and quality especially in the anterior interforaminal region as detected by CBCT and sufficient inter-arch space, minimally 12-14 mm from the ridge to the occlusal plane. The diabetic patient or patient received radiation therapy, or with parafunctional habits, and smokers should be excluded from the study.

Diagnostic and pre-operative prosthetic preparation Following the prosthetic driven implant placement protocol, all the Eligible patients already had complete dentures, their dentures were checked for adaptation, fit, stability, and occlusion. And the other patients were not wearing upper and lower complete dentures , a new denture were fabricated .

Preliminary alginate impressions (Zhermack SpA ) using a perforated stock tray were recorded, Impressions were then poured into dental stone to obtain the diagnostic model. Occlusion blocks were constructed over the diagnostic models, followed by bite registration, try-in, then the inter arch space availability for the bar was evaluated on the casts using the putty-silicon-index (Kettenbach GmbH and Co. KG ) around the artificial teeth , a minimum 13-14 mm of vertical space is required for bar-retained overdentures and finally upper and lower denture (Acrostone Dental and Medical Supplie) was delivered . Radiographic stents were fabricated as a duplicate from the fabricated patient mandibular denture with radiopaque markers (gutta percha ,Meta Dental Corp Glendale, NY ) in the centre of the teeth to guide implant positioning.

The patient was scanned CBCT while wearing the radiographic stent in the proper seating position

Surgical phase. The radiographic stent was converted to a surgical stent by drilling holes at canine areas to determine the intended surgical sites . For both groups, all patient received two implants' DENTIS Co., LTD. 3.2 x 11.5 mm (bilaterally in the canine premolar region according to bone availability in the case. All implants were placed using a surgical guide and following two-stage surgical protocol. Covering screws were screwed into the implants 3 month of healing time. In the Prosthetic stage, after 3 months of ossointegration period, the implants were exposed to receive healing collars. After two weeks, the healing collars were removed, and the soft tissue was assessed for healing. Multiunit abutments were screwed at 30 Newtons using a torque wrench. To reduce settling effect, the multiunit abutment were retightened at least two or three times at 30N torque for 10 min interval.

For both groups, primary impressions (Zhermack SpA ) were made to fabricate a special tray with window at the implant area for open tray impression technique. For impression accuracy, the long transfers coping were splinted through self-cure acrylic resin. A single-stage impression technique (putty and light body) (Kettenbach GmbH and Co. KG ) was made using silicon impression material with the open custom tray (Acrostone cold cure acrylic material; Acrostone Co).The healing caps were replaced intraorally after the impression making. Analogs were screwed over the picked-up impression coping. The final impression was poured with extra hard dental stone. (Zhermack SpA ) To assure accuracy of the master cast, acrylic verification jig (Duralay, Prestige Dentl Products, UK Ltd ) was fabricated over the impression coping using a self-cure acrylic resin. Intraoral one screw test was applied to check passivity.

Computer-generated randomization was used to divide the patients into two equal groups (1:1). An implant-retained overdenture with a cobalt-chromium bar attachment was given to Group II (the metal bar group), and Group II (the PEEK bar group) was given an overdenture with a PEEK bar attachment.

Regarding Co-Cr metal bar group, in the master cast , the multiunit abutment were attached to the implant analogues and plastic abutments were adjusted , prepared and then wax pattern coping was customized on each abutment and was connected to a preformed castable bar 2.4mm Height, (Rhein 83) The bar was placed to be away from the anterior ridge by about 2-3 mm for proper hygiene measures. The wax pattern was then sprued and casted into cobalt- chromium alloy.

Regarding PEEK bar group, the master stone cast is scanned with external desktop scanner to produce an STL (Standard Tesellation Language) file for a virtual model using the CAD/CAM software (Medit 500i.). The design of the multiunit abutment and bar (Rhein Bar )was selected from the library of the CAD software. The bar dimensions were selected according to the study bar design .

After the data acquisition, the STL file was imported to the CAM part of the CAD/CAM system to mill PEEK bar from biological high-performance polymer (Bio-HPP) (BreCAM. BioHPP, Bredent GmbH & Co.KG, Senden, Germany) block PEEK type. Multi-unit abutments were screwed to the implants and the PEEK bar was screwed to the abutments .

For all groups, Passive fit was checked visually by using a probe and by taking peri-apical radiographs to check for misfits. It was then confirmed by the one screw test which involved screwing the abutment on one side and checking the fit on the other terminal abutment.

For bar clip pickup ,all the overdentures seated and was examined intraorally, a space was made in its fitting surface that corresponded to the bar area. Condensation silicon impression material was used to block the space beneath the bar. The nylon clip (Rhein83 Italy) is firmly seated over the bar, autopolymerized acrylic resin(Acrostone cold cure acrylic material; Acrostone Co) was inserted in the relieved areas of the denture to pick up the retentive nylon clips intraorally ,the acrylic resin was set, the excess material was removed and the overdenture was delivered.

Measured outcomes Plastic clip wear and roughness were analyzed on overdenture insertion and after 3,6,9 month and 1 year of clinical usage in a 3D-surface analyzer system.27Fitting surface of denture with the nylon clip were photographed using USB Digital microscope with a built-in camera (Scope Capture Digital Microscope, Guangdong, China) connected with an IBM compatible personal computer using a fixed magnification of 120X.The images were recorded with a resolution of 1280 × 1024 pixels per image. Digital microscope images were cropped to 350 x 400 pixels using Microsoft office picture manager to standardize area of roughness measurement. WSxM software used for measure the average of heights of volumetric changes and surface roughness which expressed in μm, 28 a 3D image of the surface plastic clip was created ready for a 3-dimensional geometric analysis by the using a digital image analysis system (Image J 1.43U, National Institute of Health, USA). The intact unworn surface used as a reference.

Patients' satisfaction was evaluated After 6 month and 1 year on a scale from 1 to 10 according to the following criteria: (A) physical (stability and retention of denture), (B) Functional (chewing ability, speech ability, Pain, Comfort, Occlusion, Easiness of denture cleaning& taste of food) and(C) Aesthetic factors (Appearance of dentures & Self-image).

statistical analysis was performed with SPSS 16 ® (Statistical Package for Scientific Studies), Graph pad prism & windows excel

ELIGIBILITY:
Inclusion Criteria:

- good bone quantity and quality especially in the anterior interforaminal region as detected by CBCT and sufficient inter-arch space, minimally 12-14 mm from the ridge to the occlusal plane

Exclusion Criteria:

* diabetic patient or patient received radiation therapy, or with parafunctional habits, and smokers should be excluded from the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-08 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
attachment clip wear | base line ,3,6 and12 month
  Plastic clip wear and roughness were analyzed on overdenture insertion and after 3,6,9 month and 1 year of clinical usage in a 3D-surface analyzer system.27Fitting surface of denture with the nylon clip were photographed using USB Digital microscope with a built-in camera (Scope Capture Digital Microscope, Guangdong, China) connected with an IBM compatible personal computer using a fixed magnification of 120X.The images were recorded with a resolution of 1280 × 1024 pixels per image. Digital microscope images were cropped to 350 x 400 pixels using Microsoft office picture manager to standardize area of roughness measurement. WSxM software used for measure the average of heights of volumetric changes and surface roughness which expressed in μm, 28 a 3D image of the surface plastic clip was created ready for a 3-dimensional geometric analysis by the using a digital image analysis system (Image J 1.43U, National Institute of Health, USA). The intact unworn surface used as a reference.

SECONDARY OUTCOMES:
patient satisfaction | base line ,3,6 and12 month
  Patients' satisfaction was evaluated After 6 month and 1 year on a scale from 1 to 10 according to the following criteria: (A) physical (stability and retention of denture), (B) Functional (chewing ability, speech ability, Pain, Comfort, Occlusion, Easiness of denture cleaning& taste of food) and(C) Aesthetic factors (Appearance of dentures & Self-image).
  statistical analysis was performed with SPSS 16 ® (Statistical Package for Scientific Studies), Graph pad prism & windows excel

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Faculty of dentistry, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the data is available with the corresponding author on reasonable request